CLINICAL TRIAL: NCT06002165
Title: Testing Implementation Strategies to Support Clinic Fidelity to an Outpatient Hypertension Bundle: ACHIEVE (Advancing Community and Clinical Care for Childbirth-related Hypertension Through Implementation, Engagement, and Valuing Equity)
Brief Title: Testing Implementation Strategies to Support Clinic Fidelity to an Outpatient Hypertension Bundle
Acronym: ACHIEVE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Duke University (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-0968; OT2HL158287 (NIH)
Record Dates: First submitted 2023-08-15; First posted 2023-08-21 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy Related; Hypertension
Keywords: Hypertension; Pregnancy Related; Practice Guidelines; Prenatal Care; Quality Improvement; Implementation Science
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: The study design for the clinical trial component of the ACHIEVE initiative is a hybrid type III, multiple baseline design. Study team members will recruit and collect data from up to 20 outpatient clinics that serve pregnant patients. The clinic staff and providers will receive the intervention (a set of tailored implementation strategies) to increase their capacity to deliver timely care to patients with severe hypertension. The participating clinics will receive the intervention in three consecutive and overlapping cohorts. The first cohort, outpatient prenatal care clinics in Orange and Alamance Counties, will receive the intervention in Months 7-18 of the study. The second cohort, clinics in Durham County, will receive the intervention in Months 13-24, six months after Cohort 1 begins. The third cohort, clinics in Durham and Wake Counties, will receive the intervention in Months 19-30, twelve months after Cohort 1 begins.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Arm (Placebo Comparator): The Usual Care Arm is comprised of the clinics that are not yet receiving the intervention. All clinics participating in the study are in the Usual Care Arm until they begin the Active Implementation phase.
  Interventions: Behavioral: Usual Care
- Active Implementation Arm (Active Comparator): The Active Implementation Arm is comprised of the clinics that have started to receive the intervention, which is the ACHIEVE multi-component implementation strategy delivered by the Nurse Coordinators. All clinics (divided into 3 Cohorts) move from the Usual Care Arm into the Active Implementation Arm in sequential order (six months apart).
  Interventions: Behavioral: ACHIEVE Multi-component Implementation Strategy

INTERVENTIONS:
Behavioral: Usual Care — All clinics in North Carolina Perinatal Region IV have access to Severe HTN Bundle resources on the AIM website (https://saferbirth.org/psbs/severe-hypertension-in-pregnancy) and the locally adapted Outpatient HTN Bundle resources on the North Carolina Perinatal Region IV Provider Support Network website (https://www.mombaby.org/outpatient-bundle-for-severe-hypertension/). At baseline, the clinical leadership of all enrolled sites will receive direct communication via email that describes and provides links to the available resources. This will constitute "usual care."
  Arms: Usual Care Arm
Behavioral: ACHIEVE Multi-component Implementation Strategy — The intervention is comprised of four implementation strategies: facilitation/coaching, training, simulation, and delivering educational materials. The ACHIEVE study team, primarily the Nurse Coordinator, will engage teams within each clinic to participate in quality improvement activities utilizing these four strategies. The Nurse Coordinator will train the providers/staff on the O-HTN bundle components, facilitate corresponding office systems and workflow changes, and conduct simulations of patients with severe hypertension so care teams can practice the steps involved in recognizing and responding to episodes of severe hypertension in a timely manner.
  Arms: Active Implementation Arm

SUMMARY:
The goal of this clinical trial is to test an approach to improve care for pregnant and post-partum patients with high blood pressure. The study participants are providers and staff in prenatal care clinics, and the condition of interest is severe hypertension. The research questions are:

1. Does the ACHIEVE intervention increase the quality and accuracy of measuring patient blood pressure?
2. Does the ACHIEVE intervention increase the documentation of delivery of patient education on hypertension?
3. Does the ACHIEVE intervention result in better recognition and treatment of severe hypertension during practice sessions (simulations)?
4. Does the ACHIEVE intervention result in better recognition and treatment of severe hypertension for patients who come to the clinic?

Participants from outpatient prenatal care clinics in North Carolina will work with an ACHIEVE Nurse Coordinator who will deliver training, coaching, simulations, and educational materials. Three groups of clinics will be phased into Active Implementation every six months. The study team will examine data collected before, during, and after the intervention to see if the results show improvement.

DETAILED DESCRIPTION:
New or worsening high blood pressure in pregnancy can develop into a disease called preeclampsia. If left untreated, preeclampsia may turn into eclampsia. Eclampsia occurs when a pregnant person has a seizure or a stroke, which can lead to lifelong health problems, or even death. In 2018, 14% of pregnant people who gave birth in North Carolina experienced high blood pressure. Rural, low-income, and women of color are at greatest risk for complications of high blood pressure in pregnancy and postpartum. These same individuals also face challenges in accessing care. To improve maternal health outcomes for these patients, the Alliance for Innovation on Maternal Safety (AIM) developed the Severe Hypertension During Pregnancy and Postpartum Period Safety Bundle (HTN bundle) which includes five areas of focus: (1) Readiness of clinics to change practices (2) Recognition of high blood pressure (3) Response to patients with high blood pressure during pregnancy or postpartum; 4) Reporting/Systems Learning to track data related to clinic changes and (5) Respectful Care to ensure equity and respect in care of patients. Initially released in 2015, The HTN bundle has been used by hospitals to improve recognition and treatment of high blood pressure in birthing people. The ACHIEVE (Advancing Community and Clinical Care for Childbirth-related Hypertension through Implementation, Engagement, and Valuing Equity) Initiative was developed to support outpatient clinics in providing more effective care to pregnant individuals with high blood pressure. Adapting this bundle for community clinics providing pregnancy care has the potential to reach more birthing people outside the hospital setting who are most vulnerable to complications.

In the initial phase of ACHIEVE, the study team partnered with three rural Piedmont Health Services (PHS) clinics that serve mostly White and Latinx patients. The inpatient HTN bundle was adapted to fit their setting and re-named the Outpatient Hypertension (O-HTN) bundle. Additionally, a coalition was established to engage patients, clinic providers/staff, and the broader community to: (a) understand factors influencing maternal health including economic stability, education, health care access, and community context, (b) assess what makes it easier or harder to implement the O-HTN bundle in community outpatient clinic settings, (c) adapt the O-HTN bundle to fit those settings and populations, and (d) select and tailor changes to clinic practices using continuous cycles of learning, measuring and adapting to be the most effective and sustainable for the organization. Building on this formative work, the goal of the clinical trial is to determine the impact of four implementation strategies (training, coaching, facilitation, educational materials) in up to 20 outpatient clinics in central North Carolina. Usual clinic care for severe hypertension will be compared to the care provided after a practice has 12 months of implementation support from the ACHIEVE Nurse Coordinator. ACHIEVE partners include healthcare leadership, clinic providers and staff, community-based organizations, and individuals with lived experience who will work together on this project. If the project succeeds in improving care, the ACHIEVE model will be shared across the state and nationally to support healthier birthing people and communities.

ELIGIBILITY:
INCLUSION CRITERIA

1. Sites/Facilities Enrolling Participants

   The prenatal care clinics being recruited must meet all of the following inclusion criteria:

   a. Physical location of the clinic is in Orange, Alamance, Durham, or Wake County b. The clinic patient population includes ≥ 50 births per year c. The clinic uses an electronic health record system

   Additionally, the clinic's patient population must meet one or more of the following inclusion criteria:

   a. ≥ 50% uninsured or insured by Medicaid b. ≥ 20% Black / African American c. ≥ 20% rural residents
2. Clinic Participants

   Participants will include volunteers within the following categories:
   1. Implementation Team
   2. Care Team
   3. Medical Support Personnel
3. Patients (Patient Education Cohort)

   1. Gave birth up to six months prior to the data collection timepoint
   2. Received at least two or more prenatal care visits from the participating clinic
   3. At least one of the two prenatal care visits must occur between 20- and 34-weeks gestation
4. Patients: (Timely Delivery of Care Cohort)

   1. Pregnant or up to six weeks post-partum in the 12 months prior to the data collection timepoint.
   2. Had at least one documented episode of severe hypertension (systolic blood pressure of 160 mmHg or higher, or diastolic blood pressure of 110 mmHg or higher) during a visit encounter with a participating clinic
   3. Individual pregnant or postpartum people should have all episodes included if they present with severe range blood pressures more than once on different days

EXCLUSION CRITERIA

1. Sites/Facilities Enrolling Participants

   a. Clinics that were part of the Pilot Phase of this study b. Clinics that had recently completed a similar quality improvement project focused on severe hypertension
2. Implementation Team

   a. Provider cannot be a Medical Resident
3. Care Team

   a. Provider cannot be a Medical Resident
4. Medical Support Personnel

   a. None
5. Patients (Patient Education Cohort)

   a. None
6. Patients (Timely Delivery of Care Cohort) a. None

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Normalized percentage of achieving the highest possible score for blood pressure measurement technique | Up to 48 months
  Derived from an 11-item observation checklist with a maximum score of 11 points per observation (sample: all Medical Support Personnel who are trained to measure blood pressure for prenatal patients). The construct is fidelity to blood pressure measurement technique; a higher score represents an improvement in fidelity; the range for the checklist is 0-11 which will be translated into a normalized percentage from 0-100.
Normalized percentage of achieving the highest possible score for documentation of delivery of patient education on hypertension. | Up to 48 months
  Derived from retrospective chart audits using a chart abstraction tool and scoring system with a maximum score of 2 points per chart (sample: 20 charts per clinic randomly selected from all pregnant patients who delivered up to 6-months prior to the data collection timepoint). The construct is fidelity to the patient education protocol; a higher score represents an improvement in fidelity; the range for the score is 0-2 which will be translated into a normalized percentage from 0-100.

SECONDARY OUTCOMES:
Normalized percentage of achieving the highest possible score for recognition and response to simulated episodes of severe hypertension | Up to 13 months
  Derived from a 7-item checklist with a maximum score of 14 points per simulation (sample: all care teams in clinics that provide prenatal care.) The outcome measure will be assessed at the beginning, middle, and end of the Active Implementation phase. The construct is fidelity to recognition and response to simulated episodes of severe hypertension; a higher score represents an improvement in fidelity; the range for the checklist is 0-14 which will be translated into a normalized percentage from 0-100.
Normalized percentage of achieving the highest possible score for recognition and response to actual episodes of severe HTN | Up to 36 months
  Derived from retrospective chart audits using a chart abstraction tool and scoring system with a maximum score of 4 points per episode (sample: all episodes of severe HTN among patients who were pregnant or up to six weeks postpartum and received prenatal care from a participating clinic in the 12 months prior to the data collection timepoint). The outcome measure will be assessed in the 12 months before, during, and after the Active Implementation phase. The construct is recognition and response to actual episodes of severe hypertension; a higher score represents an improvement in fidelity; the range for the score is 0-4 which will be translated into a normalized percentage of 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Mary K Menard, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data that will be generated from our project will contain PHI. Based on ethical considerations and the need to protect the confidentiality of participants, we expect to produce the following public-use data sets to be preserved and shared:
  * Data on fidelity to protocols for Blood Pressure Measurement (observations of medical support personnel)
  * Data on fidelity to protocols for Patient Education (retrospective chart audits)
  * Data on fidelity to protocols for Recognition and Response to Episodes of Severe Hypertension (observations of care teams during simulations)
  * Data on fidelity to protocols for Recognition and Response to Episodes of Severe Hypertension (retrospective chart audits)
  Data will be aggregated at the clinic level and reported for each measurement time period. Data will include fidelity to each element of the protocol and an overall score. Clinics will be de-identified.
Supporting Information: Study Protocol, SAP
Time Frame: Publicly available data from ACHIEVE will be stored in the UNC DataVerse, a trustworthy, generalist data repository managed by theResearch Data Management Core (RDMC) at the University of North Carolina at Chapel Hill. Data will be available no more than 9 months after publication. The data will be shared and preserved for ten years, per the RDMC retention policy for UNC Dataverse.
Access Criteria: There are no anticipated factors or limitations that will affect the access, distribution or reuse of the scientific data generated by the proposal.
URL: https://dmphub.uc3prd.cdlib.net/dmps/10.48321/D17D9C08BF

REFERENCES:
- [Derived] Leeman J, Rohweder CL, Lin FC, Lightfoot AF, Costello JM, Farahi N, Harper K, Quist-Nelson J, Teal EN, Vu MB, Wheeler S, Menard MK. Community-engaged implementation of a safety bundle for pregnancy-related severe hypertension in the outpatient setting: protocol for a type 3 hybrid study with a multiple baseline design. BMC Health Serv Res. 2024 Sep 30;24(1):1156. doi: 10.1186/s12913-024-11579-8. PMID 39350133